CLINICAL TRIAL: NCT04594525
Title: Low-intensity Psychosocial Interventions in Pregnant Women in Response to COVID-19: Maternal Mental Health Matters An Interventional Study
Brief Title: Maternal Telemental Health Interventions in Response to Covid-19*
Acronym: CoronaVirus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principle investigator stopped the study as number of withdrawn participants was high so it couldnt be completed to postpartum period.
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MRC-05-087
Record Dates: First submitted 2020-10-12; First posted 2020-10-20 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-02

CONDITIONS: Perinatal Depression; Specific Phobia; Perinatal Anxiety
Keywords: Telepsychiatry; Maternal Mental Health; low-intensity psychosocial interventions
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Intervention Model Description: The design of the study: Two-arm randomized controlled trial. One Arm (Intervention): Will receive baseline assessment (personal characteristics) and standard psychological distress screening tools Plus WHO-low psychological intervention.
  One Arm (Control): baseline assessment (personal characteristics) and standard psychological distress screening tools without the WHO-low psychological intervention.
Who Masked: Outcomes Assessor
Masking Description: Blinding to data entry means a unique code will be allocated to each subject before entering the data for the analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perinatal women receiving Low intensity psychosocial interventions (Experimental): One Arm (Intervention): Will receive baseline assessment (personal characteristics) and standard psychological distress screening tools Plus WHO-low intensity psychological interventions through Telemental health.
  Interventions: Other: Low-Intensity Psychosocial Interventions through Telemental health
- Participants-Perinatal women (pregnant women and post-partum) not receiving intervention (No Intervention): One Arm (Control): baseline assessment (personal characteristics) and standard psychological distress screening tools without the WHO-low psychological intervention through Telemental health.

INTERVENTIONS:
Other: Low-Intensity Psychosocial Interventions through Telemental health — Low-Intensity Psychosocial Interventions through Telemental health (Thinking healthy): The intervention will include six sessions. Each session may last to 45 min as a max, and it will be provided through telehealth. The first session will be an introduction, while the other five sessions will be covering the period from the second pregnancy trimester to the first year of the infant's life.
  Other Names: WHO-Low intensity psychosocial Interventions
  Arms: Perinatal women receiving Low intensity psychosocial interventions

SUMMARY:
The purpose of this study is to assess the effectiveness of a telemental health intervention on the mental health of pregnant women during the COVID-19 crisis in Qatar.

DETAILED DESCRIPTION:
A list of potential participants, including contact information, will be extracted from Women Wellness and Research Center's registry. A probability sampling technique (simple random selection) will be employed to randomly select (Automated Random Number Generator) the potential participants. Then, the potential participants will be contacted and informed about the study. After consenting to participate, they will be screened for eligibility. The pregnant women who met the inclusion criteria will be enrolled and followed up until nine months after delivery. The contact details of each participant will be written on a paper and sealed in an envelope marked with either letter A or B. Upon enrolment, the participants will be randomized equally with a block size of two into two parallel arms. The pregnant women in the interventional arm will receive six sessions of a low-intensity psychosocial intervention through telemental health consultations with a trained psychologist. On the other hand, those in the control arm will not receive any intervention. The participants in both arms will be screened for psychological distress (six times) over the study period.

ELIGIBILITY:
Inclusion Criteria:

1. All pregnant women of reproductive age (18- 49) years old in the second trimester that agree and consent to receive teleconsultation.
2. No specific nationality restriction.
3. Language communicated English and Arabic.
4. Able to cooperate with data collection procedure.

Exclusion Criteria:

1. Pregnant women with psychiatric illness and following up at Sidra or HMC mental services.
2. Pregnant women receiving mental health medications (antidepressants.)
3. Cannot communicate in English or Arabic.
4. Didn't consent.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females in their Second Trimester
Enrollment: 58 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Baseline (T0) perinatal depression through the 10-points Edinburgh Postnatal Depression (Scale (EPDS-10) | Baseline in their second trimester (Beginning of 14th week till end of 27th week of gestation)
  The EPDS-10 is a validated (English and Arabic versions) instrument that assesses perinatal depression. It consists of ten questions. The total score will range from zero (no depression) to 30 (severe depression).
Change (T1-T0) from baseline perinatal depression on the 10-points Edinburgh Postnatal Depression Scale (EPDS-10) at third trimester (T1) | During the third trimester (Beginning of the 28th week till end of 42nd week of gestation)
  The EPDS-10 is a validated (English and Arabic versions) instrument that assesses perinatal depression. It consists of ten questions. The total score will range from zero (no depression) to 30 (severe depression).
Change (T2-T1) from third trimester perinatal depression on the 10-points Edinburgh Postnatal Depression Scale (EPDS-10) at 3-5 weeks postnatal (T2) | During the postnatal phase (3-5 weeks after birth)
  The EPDS-10 is a validated (English and Arabic versions) instrument that assesses perinatal depression. It consists of ten questions. The total score will range from zero (no depression) to 30 (severe depression).
Change (T3-T2) in perinatal depression on the 10-points Edinburgh Postnatal Depression Scale (EPDS-10) at 2-4 months postnatal (T3) | During the postnatal phase (2-4 months after birth)
  The EPDS-10 is a validated (English and Arabic versions) instrument that assesses perinatal depression. It consists of ten questions. The total score will range from zero (no depression) to 30 (severe depression).
Change (T4-T3) in perinatal depression on the 10-points Edinburgh Postnatal Depression Scale (EPDS-10) at 5-7 months postnatal (T4) | During the postnatal phase (5-7 months after birth)
  The EPDS-10 is a validated (English and Arabic versions) instrument that assesses perinatal depression. It consists of ten questions. The total score will range from zero (no depression) to 30 (severe depression).
Change (T5-T4) in perinatal depression on the 10-points Edinburgh Postnatal Depression Scale (EPDS-10) at 8-10 months postnatal (T5) | During the postnatal phase (8-10 months after birth)
  The EPDS-10 is a validated (English and Arabic versions) instrument that assesses perinatal depression. It consists of ten questions. The total score will range from zero (no depression) to 30 (severe depression).
Baseline (T0) Covid-19 Specific phobia through the Covid-19 Specific phobia questionnaire | Baseline in their second trimester (Beginning of 14th week till end of 27th week of gestation)
  The Covid-9 Specific phobia questionnaire consists of seven items (five-item Likert-type scale). The answers include "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree". A total score is calculated ranging from 7 to 35. The higher the score, the greater the fear of cororonavirus-19.
Change (T1-T0) in Covid-19 Specific phobia through the Covid-19 Specific phobia questionnaire at third trimester (T1) | During the third trimester (Beginning of the 28th week till end of 42nd week of gestation)
  The Covid-9 Specific phobia questionnaire consists of seven items (five-item Likert-type scale). The answers include "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree". A total score is calculated ranging from 7 to 35. The higher the score, the greater the fear of cororonavirus-19.
Change (T2-T1) in Covid-19 Specific phobia through the Covid-19 Specific phobia questionnaire at 3-5 weeks after birth (T2) | During the postnatal phase (3-5 weeks after birth)
  The Covid-9 Specific phobia questionnaire consists of seven items (five-item Likert-type scale). The answers include "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree". A total score is calculated ranging from 7 to 35. The higher the score, the greater the fear of cororonavirus-19.
Change (T3-T2) in Covid-19 Specific phobia through the Covid-19 Specific phobia questionnaire at 2-4 months after birth (T3) | During the postnatal phase (2-4 months after birth)
  The Covid-9 Specific phobia questionnaire consists of seven items (five-item Likert-type scale). The answers include "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree". A total score is calculated ranging from 7 to 35. The higher the score, the greater the fear of cororonavirus-19.
Change (T4-T3) in Covid-19 Specific phobia through the Covid-19 Specific phobia questionnaire at 5-7 months after birth (T4) | During the postnatal phase (5-7 months after birth)
  The Covid-9 Specific phobia questionnaire consists of seven items (five-item Likert-type scale). The answers include "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree". A total score is calculated ranging from 7 to 35. The higher the score, the greater the fear of cororonavirus-19.
Change (T5-T4) in Covid-19 Specific phobia through the Covid-19 Specific phobia questionnaire at 8-10 months after birth (T5) | During the postnatal phase (8-10 months after birth)
  The Covid-9 Specific phobia questionnaire consists of seven items (five-item Likert-type scale). The answers include "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree". A total score is calculated ranging from 7 to 35. The higher the score, the greater the fear of cororonavirus-19.
Baseline (T0) perinatal anxiety through a subscale of Edinburgh Postnatal Depression Scale (EPDS-3) | Baseline in their second trimester (Beginning of 14th week till end of 27th week of gestation)
  A subscale of Edinburgh Postnatal Depression Scale (EPDS-3) will be used and includes three items of EPDS-10. The total score will range from zero (no anxiety) till nine (severe anxiety).
Change (T1-T0) in perinatal anxiety through a subscale of Edinburgh Postnatal Depression Scale (EPDS-3) at third trimester (T1) | During the third trimester (Beginning of the 28th week till end of 42nd week of gestation)
  A subscale of Edinburgh Postnatal Depression Scale (EPDS-3) will be used and includes three items of EPDS-10. The total score will range from zero (no anxiety) till nine (severe anxiety).
Change (T2-T1) in perinatal anxiety through a subscale of Edinburgh Postnatal Depression Scale (EPDS-3) at 3-5 weeks after birth (T2) | During the postnatal phase (3-5 weeks after birth)
  A subscale of Edinburgh Postnatal Depression Scale (EPDS-3) will be used and includes three items of EPDS-10. The total score will range from zero (no anxiety) till nine (severe anxiety).
Change (T3-T2) in perinatal anxiety through a subscale of Edinburgh Postnatal Depression Scale (EPDS-3) at 2-4 months after birth (T3) | During the postnatal phase (2-4 months after birth)
  A subscale of Edinburgh Postnatal Depression Scale (EPDS-3) will be used and includes three items of EPDS-10. The total score will range from zero (no anxiety) till nine (severe anxiety).
Change (T4-T3) in perinatal anxiety through a subscale of Edinburgh Postnatal Depression Scale (EPDS-3) at 5-7 months after birth (T4) | During the postnatal phase (5-7 months after birth)
  A subscale of Edinburgh Postnatal Depression Scale (EPDS-3) will be used and includes three items of EPDS-10. The total score will range from zero (no anxiety) till nine (severe anxiety).
Change (T5-T4) in perinatal anxiety through a subscale of Edinburgh Postnatal Depression Scale (EPDS-3) at 8-10 months after birth (T5) | During the postnatal phase (8-10 months after birth)
  A subscale of Edinburgh Postnatal Depression Scale (EPDS-3) will be used and includes three items of EPDS-10. The total score will range from zero (no anxiety) till nine (severe anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- HMC, Doha, Qatar

REFERENCES:
- [Derived] Naja S, Elyamani R, Chehab M, Ali Siddig Ahmed M, Babeker G, Lawand G, Singh R, Adli N, Mohamad T, Bougmiza I. The impact of telemental health interventions on maternal mental health outcomes: a pilot randomized controlled trial during the COVID-19 pandemic. Health Psychol Behav Med. 2022 Dec 28;11(1):1-21. doi: 10.1080/21642850.2022.2155167. eCollection 2023. PMID 36606005
- [Derived] Naja S, Elyamani R, Chehab M, Siddig M, Al Ibrahim A, Mohamad T, Singh R, Bougmiza I. Maternal low-intensity psychosocial telemental interventions in response to COVID-19 in Qatar: study protocol for a randomized controlled trial. Trials. 2021 Jun 7;22(1):382. doi: 10.1186/s13063-021-05339-w. PMID 34099007